CLINICAL TRIAL: NCT03395912
Title: Efficacy of a Single-shot Wound Infiltration With Bupivacaine/Adrenalin During Cesarean Section in Reducing Postoperative Pain. A Randomized Prospective Controlled Trial
Brief Title: Wound Infiltration With Bupivacaine/Adrenalin During Cesarean Section and Postoperative Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0151-17-EMC
Record Dates: First submitted 2017-12-21; First posted 2018-01-10 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Cesarean Section
Keywords: local anesthetics infiltration; cesarean section pain relief
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Infiltration of the subcutaneous layer with local anesthetic and combined with adrenaline.
  Interventions: Drug: Intervention
- control (No Intervention): Abdominal layers will be closed without Infiltration .

INTERVENTIONS:
Drug: Intervention — After closing the fascia above the rectus muscles, and before closing the skin, the subcutaneous layer will be infiltrated on both sides of the incision (top and bottom) by 30 ml of 0.25% BUPIVACAINE and ADRENALIN at 1: 200,000 concentration and then closing the skin.
  Other Names: local anesthetic infiltration
  Arms: Intervention

SUMMARY:
Thus study evaluates the advantage of infiltration of the surgical wound by local anesthetics in cesarean section on post operative pain relief. In the study group before closing the skin, both sides of the incision (top and bottom) will be infiltrated by 30 ml of 0.25% BUPIVACAINE and ADRENALIN at 1: 200,000 concentration and then closing the skin. In the control group, the skin will be closed without infiltration. Our hypothesis is that subcutaneous infiltration of the surgical wound by BUPIVACAINE + ADRENALIN at the end of cesarean section will reduce the intensity of post operative pain.

DETAILED DESCRIPTION:
Cesarean section is one of the most common procedures in the world. There is an advantage in preventing pain after cesarean section, as opposed to treating pain that has already started. The infiltration of surgical wounds by local anesthetics is accepted as an effective method for preventing pain after various operations. In this study women who are admitted for a cesarean section will be randomly allocated into 2 groups. In the study group after the closure of the fascia above the rectus muscles, and before closing the skin, both sides of the incision (top and bottom) will be infiltrated by 30 ml of 0.25% BUPIVACAINE and ADRENALIN at 1: 200,000 concentration and then closing the skin. In the control group, the skin will be closed without infiltration.

ELIGIBILITY:
Inclusion Criteria:

* cesarean section with regional anesthesia
* singleton
* pfannenstiel incision

Exclusion Criteria:

* cesarean section with general anesthesia
* maternal liver or kidney disease
* allergy to Bupivacaine
* allergy to Adrenalin
* intrauterine fetal death
* major fetal malformations

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Self reported pain intensity upon receipt of a woman after cesarean section to the maternity department. | up to 24 hours
  Visual analogue scale pain severity with scale from 0 to 10, with score 10 representing the maximum level of pain.

SECONDARY OUTCOMES:
Length of the cesarean section | up to 24 hours
  Time from first incision to the end of incision closure
Time from surgery to mobility | up to 48 hours
  Time from the end of surgery to mobility
Time from surgery to breastfeeding | up to 4 days
  Time from the end of surgery to breastfeeding
Need for opioids | up to 4 days
  Type and dosage of opioids needed
Surgical site hematoma | 4 days
  Post operative surgical site hematoma
surgical site infection | up to 42 days
  Post operative surgical site infection
questionnaire | up to 4 days
  Post operative women's satisfaction with scale from 0 to 10, with score 10 representing the maximum level of satisfaction.
Length of stay from surgery to discharge | up to 4 days
  Length of stay from surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Gali Garmi, MD, Principal Investigator — HaEmek Medical Center, Afula, Israel
Locations (1):
- HaEmek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Karlstrom A, Engstrom-Olofsson R, Norbergh KG, Sjoling M, Hildingsson I. Postoperative pain after cesarean birth affects breastfeeding and infant care. J Obstet Gynecol Neonatal Nurs. 2007 Sep-Oct;36(5):430-40. doi: 10.1111/j.1552-6909.2007.00160.x. PMID 17880313
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Yefet E, Taha H, Salim R, Hasanein J, Carmeli Y, Schwartz N, Nachum Z. Fixed time interval compared with on-demand oral analgesia protocols for post-caesarean pain: a randomised controlled trial. BJOG. 2017 Jun;124(7):1063-1070. doi: 10.1111/1471-0528.14546. Epub 2017 Feb 25. PMID 28236348
- [Result] Adesope O, Ituk U, Habib AS. Local anaesthetic wound infiltration for postcaesarean section analgesia: A systematic review and meta-analysis. Eur J Anaesthesiol. 2016 Oct;33(10):731-42. doi: 10.1097/EJA.0000000000000462. PMID 27259092
- [Result] Fredman B, Shapiro A, Zohar E, Feldman E, Shorer S, Rawal N, Jedeikin R. The analgesic efficacy of patient-controlled ropivacaine instillation after Cesarean delivery. Anesth Analg. 2000 Dec;91(6):1436-40. doi: 10.1097/00000539-200012000-00025. PMID 11093995
- [Result] Givens VA, Lipscomb GH, Meyer NL. A randomized trial of postoperative wound irrigation with local anesthetic for pain after cesarean delivery. Am J Obstet Gynecol. 2002 Jun;186(6):1188-91. doi: 10.1067/mob.2002.122984. PMID 12066096
- [Result] Lavand'homme PM, Roelants F, Waterloos H, De Kock MF. Postoperative analgesic effects of continuous wound infiltration with diclofenac after elective cesarean delivery. Anesthesiology. 2007 Jun;106(6):1220-5. doi: 10.1097/01.anes.0000267606.17387.1d. PMID 17525598
- [Result] Mecklem DW, Humphrey MD, Hicks RW. Efficacy of bupivacaine delivered by wound catheter for post-Caesarean section analgesia. Aust N Z J Obstet Gynaecol. 1995 Nov;35(4):416-21. doi: 10.1111/j.1479-828x.1995.tb02156.x. PMID 8717568
- [Result] Tuncer S, Aysolmaz G, Reisli R, Erol A, Yalcin N, Yosunkaya A. [The effects of the administration of subfacial levobupivacaine infusion with the ON-Q pain pump system on postoperative analgesia and tramadol consumption in cesarean operations]. Agri. 2010 Apr;22(2):73-8. Turkish. PMID 20582749
- [Result] Zohar E, Shapiro A, Eidinov A, Fishman A, Fredman B. Postcesarean analgesia: the efficacy of bupivacaine wound instillation with and without supplemental diclofenac. J Clin Anesth. 2006 Sep;18(6):415-21. doi: 10.1016/j.jclinane.2006.01.001. PMID 16980157
- [Result] Jolly C, Jathieres F, Keita H, Jaouen E, Guyot B, Torre A. Cesarean analgesia using levobupivacaine continuous wound infiltration: a randomized trial. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:125-30. doi: 10.1016/j.ejogrb.2015.08.023. Epub 2015 Aug 25. PMID 26366789
- [Result] Corsini T, Cuvillon P, Forgeot A, Chapelle C, Seffert P, Chauleur C. [Single-dose intraincisional levobupivacaine infiltration in caesarean postoperative analgesia: a placebo-controlled double-blind randomized trial]. Ann Fr Anesth Reanim. 2013 Jan;32(1):25-30. doi: 10.1016/j.annfar.2012.10.035. Epub 2012 Dec 21. French. PMID 23260628
- [Result] Ducarme G, Sillou S, Wernet A, Davitian C, Poujade O, Ceccaldi PF, Bougeois B, Luton D. [Single-shot ropivacaine wound infiltration during cesarean section for postoperative pain relief]. Gynecol Obstet Fertil. 2012 Jan;40(1):10-3. doi: 10.1016/j.gyobfe.2011.07.035. Epub 2011 Oct 22. French. PMID 22024157
- [Result] Bensghir M, Elwali A, Miller C, Azendour H, Drissi M, Bakkali H, Belyamani L, Atmani M, Drissi Kamili N. [Effects of skin infiltration with ropivacaine 0,75% on postoperative pain after caesarean section]. Gynecol Obstet Fertil. 2008 May;36(5):516-20. doi: 10.1016/j.gyobfe.2008.03.007. Epub 2008 May 7. French. PMID 18467147
- [Result] Pavy T, Gambling D, Kliffer P, Munro A, Merrick PM, Douglas J. Effect of preoperative skin infiltration with 0.5% bupivacaine on postoperative pain following cesarean section under spinal anesthesia. Int J Obstet Anesth. 1994 Oct;3(4):199-202. doi: 10.1016/0959-289x(94)90068-x. PMID 15636950
- [Result] Sekhavat L, Behdad S. Preoperative analgesia with local lidocaine for cesarean delivery pain relief. J Matern Fetal Neonatal Med. 2011 Jul;24(7):891-3. doi: 10.3109/14767058.2010.537410. Epub 2011 Jan 10. PMID 21219106
- [Result] Trotter TN, Hayes-Gregson P, Robinson S, Cole L, Coley S, Fell D. Wound infiltration of local anaesthetic after lower segment caesarean section. Anaesthesia. 1991 May;46(5):404-7. doi: 10.1111/j.1365-2044.1991.tb09558.x. PMID 2035794
- [Result] Parascandola SA, Ibanez J, Keir G, Anderson J, Plankey M, Flynn D, Cody C, De Marchi L, Margolis M, Blair Marshall M. Liposomal bupivacaine versus bupivacaine/epinephrine after video-assisted thoracoscopic wedge resectiondagger. Interact Cardiovasc Thorac Surg. 2017 Jun 1;24(6):925-930. doi: 10.1093/icvts/ivx044. PMID 28329326
- [Result] Metaxotos NG, Asplund O, Hayes M. The efficacy of bupivacaine with adrenaline in reducing pain and bleeding associated with breast reduction: a prospective trial. Br J Plast Surg. 1999 Jun;52(4):290-3. doi: 10.1054/bjps.1998.0129. PMID 10624296
- [Result] Li X, Zhou M, Shi X, Yang H, Li Y, Li J, Yang M, Yuan H. Local anaesthetic wound infiltration used for caesarean section pain relief: a meta-analysis. Int J Clin Exp Med. 2015 Jun 15;8(6):10213-24. eCollection 2015. PMID 26309720
- [Derived] Garmi G, Parasol M, Zafran N, Rudin M, Romano S, Salim R. Efficacy of Single Wound Infiltration With Bupivacaine and Adrenaline During Cesarean Delivery for Reduction of Postoperative Pain: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2242203. doi: 10.1001/jamanetworkopen.2022.42203. PMID 36378307